CLINICAL TRIAL: NCT04330105
Title: Subclinical Cardiac Involvement in Patients With Inflamatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hossam Eldin Mohammed Essam Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Hossam Eldin Mohammed Essam Abdelhafez, Subclinical cardiac involvement in patients with inflamatory bowel disease, Assiut University
Organization: Assiut University (Other)
Other Study IDs: inflamatory bowel disease
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ECG, HolterECG ,Echocardiography — ECG, HolterECG ,Echocardiography to determine any type of arrythmia,ischaemic heart disease,valvular heart disease,systolic and diastolic dysfunction

SUMMARY:
Aim of the study is to determine the prevelance of subclinical cardiac involvement in patients with inflamatory bowel disease.

DETAILED DESCRIPTION:
Cardiovascular manifestations in patients with IBD mostly occur as immune-related consequences and include the following: pericarditis, myocarditis, venous and arterial thromboembolism, left ventricle impairment, arrhythmias and conduction disorders and valvulopathy .

The prevalence of classical cardiovascular risk factors is relatively lower in IBD patients than in the general population . However, the risk of coronary heart disease is higher in IBD patients .

The pathophysiology of cardiac involvement may be Systemic inflammation for prolonged periods that can cause platelet aggregation and endothelial dysfunction leading to the development of atherosclerosis and CVD .

The chronic inflammatory condition found in IBD is the key element in the pathogenesis of arrhythmias.

In IBD, inflammation causes mitral and aortic valvulopathies , excess TNF-α causes the thickening and shortening of the leaflets, resulting in regurgitation .

Medications of IBD may be involved in pathogenesis of cardiac involvement as follows 5-ASA and its derivatives can cause myopericarditis . Atrial fibrillation and prolonged QT interval may occur during azathioprine use .

Cyclosporine is associated with increased risk of hypertension, arrhythmias, acute coronary syndrome, and heart failure .

Biological molecules are associated with increased arrhythmogenic risks . Primary preventive measures of arterial thromboembolism include maintaining the remission, strict control of cardiovascular risk factors .

The diagnostic modalities to find out cardiac involvement include; The 12-lead electrocardiogram . Transthoracic echocardiography which represent the method of choice to evaluate both systolic and diastolic functions of Lt ventricle.

Methodology:

All Patints will be subjected to the followings :

Full history taking including

* Duration of illness
* Symptoms of disease activity
* Symptoms of extraintestinal manifestation
* Family history of cardiac disease
* History of traditional cardiovascular risk factors diabetes,hypertension,Dyslipidaemia,cigarette smooking)
* Therapeutic history Examination
* Body mass index.
* Vital signs( pulse,blood pressure,temperature).
* Cardiac examination.

Labaratory investigations

* Complete blood count - serum electrolytes
* ESR - CRP
* lipid profile - blood glucose level
* TSH,T3,T4

ECG

* Ischaemic changes
* Any type of arrythmia
* Prolonged QT interaval

Holter ECG

Echocardiography

* Systolic and diastolic dysfunctions
* Wall motion abnormalities
* Valvular heart disease
* Ventricular hypertrophy
* Atrial and ventricular dimentions

ELIGIBILITY:
Inclusion Criteria:

* Inflamatory bowel disease patients without previous history of cardiac disease.

Exclusion Criteria:

* Patients known to have previous cardiac disease.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: IBD patients who have no previous history of cardiac disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
determine the prevelance of cardiac involvement in inflamatory bowel disease | Baseline
  Assesment of cardiac involvement in inflamatory bowel disease byECG,HolterECG andEchocardiography